CLINICAL TRIAL: NCT06198062
Title: Effects of Paraffin Wax Bath Therapy With and Without Muscle Energy Technique in Children With Post Burn Hand Contracture
Brief Title: Effects of Paraffin Wax Therapy vs METs in Post Burn Hand Contractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0736
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Contracture, Hand
Keywords: Paraffin wax; METS; Contracture; Burn
MeSH Terms: conditions — Contracture; Burns

STUDY DESIGN:
Intervention Model Description: This will be randomized control trail to see effects of Paraffin wax bath therapy with and without muscle energy technique in children with post burn hand contracture
Who Masked: Participant
Masking Description: Participants will get a separate treatment protocol and possible efforts will be mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin wax bath therapy (Experimental): Heat therapy for the relief of joint pain and stiffness was established using paraffin and prolonged stretching. When used as a treatment method, paraffin wax is heated to a temperature between 115 and 118 degrees. One step of the paraffin treatment is cleaning. (1) Drying the damaged area and making sure the skin is covered in plastic, (2) Wrapping any small open wounds in plastic, (3) Applying paraffin wax to the affected area, (4) Stretching the affected extremity for 20 minutes, (5)Covering the area with an ACE bandage or a towel to prevent the wax from cooling too quickly
  Interventions: Other: Paraffin wax bath therapy
- Muscle energy technique (Experimental): Reciprocal inhibition, hypertonic antagonists can reflexively inhibiting their agonist muscle. Therefore, in the presence of short and tight antagonist muscles, restoring normal muscle tone and length should be first addressed. MET involves the subject to voluntarily contract the muscle in a precisely controlled direction against the therapist's counter force. Its therapeutic effects are to reduce pain, reduce muscle tone, stretch tightened muscles, strengthen the weak muscles, improve local circulation and mobilize joint restrictions. Anatomical structures that contribute to stiffness at the joint states that the joint capsule, surrounding inter-muscular fasciae and muscles, tendons and skin tissue account for restriction at the joint. Relaxation of the antagonist muscle occurs due to actively contracting the agonist muscle
  Interventions: Other: Paraffin Wax Bath Therapy and Muscle Energy Techniques

INTERVENTIONS:
Other: Paraffin wax bath therapy — this group receive paraffin wax. Each session will last between 40 and 50 min, 2 sessions per week, for total 6 weeks
  Arms: Paraffin wax bath therapy
Other: Paraffin Wax Bath Therapy and Muscle Energy Techniques — This group receive paraffin wax bath therapy along with muscle energy techniques. Each session will be conducted for 40 to 50 mins, 3 sessions in a week for total 6 weeks
  Arms: Muscle energy technique

SUMMARY:
The degree of the burn and the rate of scar development during healing are the main determinants of loss of hand function following thermal injury. Compared to adults, managing these injuries in children presents unique challenges due to three factors: (I) children's thin hand skin makes it difficult to protect deep hilar structures; (II) rapid growth of the hand and fingers in the second and third years of life can cause contusion scar deformity; and (III) treatment is frequently challenging due to the young child's lack of cooperation. The manual technique known as Muscle Energy Technique (MET) primarily targets the soft tissues, although it also has significant effects on the muscles. Osteopaths and is currently utilized by a variety of manual therapy professions as a contribution to joint mobilization. This method is also known as the active muscular relaxation technique or the muscle energy technique. Exercise is necessary to maintain mobility, which in turn depends on overcoming dryness and decreased suppleness of the scar tissue across the joint, which in turn depends on preventing joint stiffness. Heat therapy for the relief of joint pain and stiffness was established using paraffin and prolonged stretching. When used as a treatment method, paraffin wax is heated to a temperature between 115 and 118 degrees.

DETAILED DESCRIPTION:
The degree of the burn and the rate of scar development during healing are the main determinants of loss of hand function following thermal injury. Compared to adults, managing these injuries in children presents unique challenges due to three factors: (I) children's thin hand skin makes it difficult to protect deep hilar structures; (II) rapid growth of the hand and fingers in the second and third years of life can cause contusion scar deformity; and (III) treatment is frequently challenging due to the young child's lack of cooperation. The manual technique known as Muscle Energy Technique (MET) primarily targets the soft tissues, although it also has significant effects on the muscles. Osteopaths and is currently utilized by a variety of manual therapy professions as a contribution to joint mobilization. This method is also known as the active muscular relaxation technique or the muscle energy technique. Exercise is necessary to maintain mobility, which in turn depends on overcoming dryness and decreased suppleness of the scar tissue across the joint, which in turn depends on preventing joint stiffness. Heat therapy for the relief of joint pain and stiffness was established using paraffin and prolonged stretching. When used as a treatment method, paraffin wax is heated to a temperature between 115 and 118 degrees.

It will be randomized controlled trail. In which convenient sampling technique will be used. Two groups will be formed in which participants will be divided by lottery method. Group A will be treated by paraffin wax bath therapy and Group B treated by paraffin wax bath therapy with muscle energy technique. The result after statistical analysis will either show this intervention is effective or not. Result will be analyzed on SPSS

ELIGIBILITY:
Inclusion Criteria

* Child with age 4 to 12 yrs
* Mild and moderate type of contracture
* Loss up to one third and two third of ranges
* Recently healed wounds to be sure that no open area exist
* Post burn contracture
* Without fragile blistering

Exclusion Criteria

* Severe type of contractures
* Loss of more than two-third of ranges
* Any spinal cord injuries
* Children with rigid spastic contractures
* Contractures other than burn
* Wounds that have open area and risk of bleeding occurs

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Goniometer | 6 weeks
  Measuring a joint angle with a universal goniometer has moderate to excellent reliability. It can therefore, be used as a repeatable device for measuring the range of motion of the joint. According to an article the inter-tester reliability of goniometer is 0.98 and ICC is 0.99 and validity 0.97-0.98. The results of this study indicates that goniometric measurement are both valid and reliable.
ABILHAND-kids Questionnaires | 6 weeks
  ABILHAND-Kids is use to measure the manual ability of hand in children. The scale used for face to face interview of the parents of the child. The interview will be conduct twice. On the first visit and after an interval of 15 days. The scale consist of different activities parents are asked to fill the questionnaire by estimating their child difficulty on three levels.
  Impossible: the child is unable to perform the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Aiman Arif, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riaz HM, Ashraf Cheema S. Paraffin wax bath therapy versus therapeutic ultrasound in management of post burn contractures of small joints of hand. Int J Burns Trauma. 2021 Jun 15;11(3):245-250. eCollection 2021. PMID 34336391